CLINICAL TRIAL: NCT01811199
Title: Dexamethasone Reduces Postoperative Emesis by Decreasing PGF2α and LTC4 Levels
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, A.Ozdemir Aktan, professor of surgery, Marmara University
Other Study IDs: 09.2011.0024
Record Dates: First submitted 2013-03-06; First posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Thyroid Cancer; Breast Cancer
Keywords: Thyroid cancer; Breast cancer; Dexamethasone; Emesis
MeSH Terms: conditions — Thyroid Neoplasms; Breast Neoplasms; Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: Dexamethasone reduces postoperative emesis in thyroidectomy and mastectomy patients.

DETAILED DESCRIPTION:
This study has been done to further study the effectiveness of dexamethasone in the prevention of postoperative emesis after breast and thyroid surgery and at the same time, the mechanism of action was investigated. In this prospective, randomized controlled trial it was hypothesized that corticosteroids exert their antiemetic effects in postoperative period via plasma prostaglandin F2 alpha (PGF2 α) and plasma leukotriene C4 (LTC4) inhibition.

ELIGIBILITY:
Inclusion Criteria:

* breast and thyroid cancer patients no neoadjuvant treated no NSAID or steroid usage heallthy volunteers, signed the informed consent

Exclusion Criteria:

* ones who did not sign the consent form NSAID or steroid users

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thyroidectomy and mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-04 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants will be evaluated to show effect of dexamethasone in reducing postoperative emesis | up to 3 days
  participants will be followed for the duration of hospital stay, till they are discharged in avarage 3 days for postoperative emesis.

CONTACTS AND LOCATIONS:
Overall Officials: A.Ozdemir Aktan, MD,prof, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)